CLINICAL TRIAL: NCT06828484
Title: Evaluating the Clinical and Biological Response of an Acetone-Precipitated Cat Hair Allergen Extract (AP Cat) in a Nasal Allergen Challenge (NAC).
Brief Title: Allergenic Extract Standardized Cat Hair AP in an Allergic Rhinitis Model.
Acronym: AP-CAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Anne Ellis, Principal Investigator, Queen's University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AP-CAT
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Allergic Rhinitis
Keywords: Allergy; Allergic Rhinitis; Perennial Allergies; Cat Allergies; Allergen Exposure Models; Nasal Allergen Challenge
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Both allergic (Arm 1) and non-allergic (Arm 2) groups will receive the same intervention (AP Cat) through the NAC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allergic Participant AP-Cat Challenge (Experimental)
  Interventions: Drug: Allergenic Extract Standardized Cat Hair Acetone-Precipitated (AP)
- Non-Allergic Participant AP-Cat Challenge (Experimental)
  Interventions: Drug: Allergenic Extract Standardized Cat Hair Acetone-Precipitated (AP)

INTERVENTIONS:
Drug: Allergenic Extract Standardized Cat Hair Acetone-Precipitated (AP) — Cat-allergic and non-allergic participants will be exposed to AP Cat in the NAC.
  Other Names: AP Cat

SUMMARY:
The goal of this study is to learn if a cat allergen extract known as Allergenic Extract Standardized Cat Hair Acetone Precipitated (AP Cat) can induce allergic rhinitis (AR) in a nasal allergen challenge model in cat-allergic people. The main questions this study aims to answer are:

1. Does AP Cat induce nasal symptoms of allergic rhinitis in cat-allergic participants when delivered intranasally?
2. Does AP Cat reduce elements in the blood and nose that are known to be associated with allergies?

Both allergic and non-allergic participants will be recruited into this study.

Allergic participants will:

* Be challenged with AP Cat via the Nasal Allergen Challenge (NAC), which involves administration of this allergen extract directly into the nose.
* Have nasal fluid and blood samples collected at various timepoints up to 24 hours after exposure to the allergen in the NAC.
* Visit the study site three separate times:

  1. At screening (Visit 1), to determine eligibility to participate in this study
  2. At the baseline NAC visit (Visit 2)
  3. At the 24-hour post-NAC follow-up visit (Visit 3)
* Complete nasal symptom questionnaires.
* Complete a questionnaire about their regular exposure to cats.

Non-allergic participants will:

* Be challenged with AP Cat via the NAC, which involves administration of this allergen extract directly into the nose.
* Have nasal fluid and blood samples collected at various timepoints up to 24 hours after exposure to the allergen in the NAC.
* Visit the study site three separate times:

  1. At screening (Visit 1), to determine eligibility to participate in this study
  2. At the baseline NAC visit (Visit 2)
  3. At the 24-hour post-NAC follow-up visit (Visit 3)
* Complete nasal symptom questionnaires.

This study will compare the nasal symptoms and allergic markers collected from the nasal fluid and blood samples between allergic and non-allergic participants at baseline and various timepoints post-NAC exposure.

DETAILED DESCRIPTION:
The purpose of this single-centre prospective cohort study is to evaluate the use of AP Cat in the NAC. Allergen extracts are used in skin prick testing, allergy research, and immunotherapy. AP Cat is a new formulation of a cat allergen extract approved for use in skin prick testing, but has not yet been studied in the NAC.

This study will enrol non-pregnant and non-lactating female and/or male participants. 15 cat-allergic participants and 5 non-allergic participants from 18-70 years old will be recruited from the Kingston, Frontenac, Lennox, and Addington region in Ontario, Canada. All 20 participants will attend three study visits: Visit 1 (Screening Visit), Visit 2 (NAC Exposure Visit), and Visit 3 (Follow-up Visit). Visit 2 will occur at least 21 days after Visit 1. Visit 3 will occur 24 hours after the onset of the NAC during visit 2. At each visit, symptom scores, nasal fluid samples, and blood samples will be collected.

The investigators hypothesize that AP Cat will induce AR-related outcomes (Total Nasal Symptom Score (TNSS), Peak Nasal Inspiratory Flow (PNIF), Total Ocular Symptom Score (TOSS), Total Rhinoconjunctivitis Symptom Score (TRSS)) in cat-allergic participants after exposure in the NAC. The investigators also hypothesize that AP Cat will increase the release of allergic mediators (Interleukin-4 (IL4),IL-5, IL-10, IL-13, Eotaxin-1, Monocyte Chemoattractant Protein-1 (MCP-1), Macrophage Inflammatory Protein-1 Beta (MIP-1β), and alarmins (IL-17E/IL-25, IL-33)) in cat-allergic participants after the NAC. Additionally, the investigators expect that nasal white blood cell counts and peripheral total immunoglobulin E (tIgE) levels will increase in cat-allergic participants after the NAC. Furthermore, the investigators hypothesize that no significant changes to nasal symptoms, allergic mediator levels, nasal eosinophil counts, or tIgE levels will occur in the non-allergic participants, which serve as controls.

ELIGIBILITY:
Inclusion Criteria:

To be considered for inclusion in this study, all participants must be:

* A healthy, ambulatory male, female, or intersex volunteer between the ages of 18 to 70 years of age.
* Able to understand and willing to provide written informed consent.
* Able and willing to comply with study requirements.

To be enrolled as an allergic participant, participants must:

* Have a minimum 2-year history of AR symptoms upon exposure to cats.
* Have a positive skin prick response to AP cat allergen, defined as a wheal diameter ≥ 5 mm compared to the negative control wheal. This result must be achieved at visit 1.
* Have a TNSS of greater than or equal to 8/12 and at least a 50% drop in PNIF in response to the allergen titration challenge at visit 1.

To be enrolled as a non-allergic participant, participants must:

* Produce a negative skin test response to a panel of relevant aeroallergens tested at visit 1 or within 12 months before visit 1 at the research site.
* Produce a negative Nasal Allergen Challenge, defined by a TNSS response of less than 4/12 and a PNIF reduction of less than or equal to 20% after 10 minutes in response to the highest allergen concentration at visit 1.

Exclusion Criteria:

* Participant has abnormalities detected on physical examination considered by the investigator to be clinically significant.
* Participant has a history of any disease or disorder that, in the judgement of the investigator, would impact the participant's safety or the results of the study.
* Participant has a significant history of alcohol or drug abuse in the judgment of the Principal Investigator or delegate.
* Participant is pregnant, lactating, or actively trying to become pregnant.
* Participant is unable to comply with the washout periods for restricted medications.
* Participant has signs/symptoms of active seasonal AR or is allergic to a seasonal allergen that is present in the outdoor environment during visit 1 and visit 2 and which the Principal Investigator judges would impact the outcome of the study.
* Participant has any structural nasal abnormalities or nasal polyps on examination or a history of frequent nose bleeding, as determined by a nasal examination at screening and prior to the NAC, in the judgement of the principal investigator.
* Participant has undergone nasal surgery within the previous 3 months before visit 1.
* Participant has experienced an upper or lower respiratory infection within 2 weeks prior to the NAC visit.
* Participant exhibits any signs or symptoms of a respiratory infection prior to any visit, as per Principal Investigator judgement.
* Participant reports a TNSS of greater than or equal to 4 prior to the titration challenge at visit 1 or immediately prior to allergen challenge at visit 2, as per Principal Investigator judgement.
* Participant reports a TNSS change of greater than 2 from baseline, after the diluent challenge at visit 1.
* Participants with asthma requiring the use of a short-acting beta agonist greater than twice a week (unless for viral asthma) or with severe asthma requiring maintenance high doses of inhaled or oral corticosteroids or biologic therapy (Omalizumab/Mepolizumab/Resilizumab).
* Participant has a history of cat allergen induced asthma, unless well controlled on low-dose inhaled corticosteroids or PRN inhaled corticosteroid/long-acting beta-agonist as per Principal Investigator discretion.
* Participant is currently receiving cat allergen specific immunotherapy or concluded a course of cat immunotherapy in the last 3 years.
* Participant has a history of positive test results for HIV, Tuberculosis (not due to vaccination), Hepatitis B (not due to vaccination) or Hepatitis C.
* Participant has received an investigational product within the previous 30 days.
* Participant is unable and/or unlikely to comprehend and/or follow the protocol over the duration of the study. Participant is unwilling to attend study visits or adhere to the study protocol, in the judgement of the Principal investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Pre-NAC up to 24 hours post-NAC.
  To evaluate the effect of NAC exposure to AP Cat on TNSS (where a score of 0 indicates no nasal allergic symptoms while a score of 12 indicates the maximum nasal symptoms) compared to baseline measures in cat-allergic participants.

SECONDARY OUTCOMES:
Peak Nasal Inspiratory Flow (PNIF) | Pre-NAC up to 24 hours post-NAC.
  To evaluate the effect of NAC exposure to AP Cat on PNIF compared to baseline measures in cat-allergic participants.
Total Ocular Symptom Score (TOSS) | Pre-NAC up to 24 hours post-NAC.
  To evaluate the effect of NAC exposure to AP Cat on TOSS (where a score of 0 indicates no ocular symptoms whereas a score of 9 indicates maximum ocular symptoms) compared to baseline measures in cat-allergic participants.
Total Rhinoconjunctivitis Symptom Score (TRSS) | Pre-NAC up to 24 hours post-NAC.
  To evaluate the effect of NAC exposure to AP Cat on TRSS (where a score of 0 indicates no rhinoconjunctivitis symptoms whereas a score of 24 indicates maximum rhinoconjunctivitis symptoms) compared to baseline measures in cat-allergic participants.
Safety Outcome Scoring | From enrolment to the final study visit.
  To evaluate the safety of NAC exposure to Allergenic Extract Standardized Cat Hair AP (coughing, wheezing, chest tightness, shortness of breath, where a score of 0 indicates no symptoms whereas a score of 12 indicates maximum symptoms).
Concentration of alarmins (IL-17E/IL-25, IL-33) from serum. | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the effect of using AP Cat in an NAC on peripheral allergic biomarkers pre- and post-NAC.
Concentration of alarmins (IL-17E/IL-25, IL-33) from nasal fluid. | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the effect of using AP Cat in an NAC on nasal allergic biomarkers pre- and post-NAC.
Concentration of type 2 cytokines (IL-4, IL-5, IL-10, IL-13) from serum. | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the effect of using AP Cat in an NAC on peripheral allergic biomarkers pre- and post-NAC.
Concentration of type 2 cytokines (IL-4, IL-5, IL-10, IL-13) from nasal fluid. | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the effect of using AP Cat in an NAC on nasal allergic biomarkers pre- and post-NAC.
Concentration of chemokines (Eotaxin-1, MCP-1, MIP-1B) from serum. | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the effect of using AP Cat in an NAC on peripheral allergic biomarkers pre- and post-NAC.
Concentration of chemokines (Eotaxin-1, MCP-1, MIP-1B) from nasal fluid. | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the effect of using AP Cat in an NAC on nasal allergic biomarkers pre- and post-NAC.
Concentration of total immunoglobulin E from serum. | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the effect of using AP Cat in an NAC on peripheral biomarkers pre- and post-NAC.
White blood cell count from nasal lavage. | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the effect of using AP Cat in an NAC on nasal allergic biomarkers pre- and post-NAC.

OTHER OUTCOMES:
Skin Prick Test Wheal Diameter | Screening, baseline, 3 hours post-NAC, 6 hours post-NAC, 24 hours post-NAC.
  To evaluate the use of AP Cat in skin prick testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre - Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No